CLINICAL TRIAL: NCT04855864
Title: Better Functional Outcome When Preserving, Substituting or Sacrificing ACL During TKA? A Prospective Functional Analysis of a Bicruciate Retaining, a Bicruciate Stabilized and a Posterior Stabilized Prosthetic Design
Brief Title: Journey Bicruciate Stabilized (BCS) Design and Legion Posterior Stabilized (PS) Design; Comparative Study
Acronym: BCR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: S64561
Record Dates: First submitted 2021-04-16; First posted 2021-04-22 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Primary Total Knee Arthroplasty
Keywords: Journey BCS®; Journey XR®; Legion PS®

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BCR TKA (Other): Patients with intact and functional ACL and PCL will be treated with the BCR design
  Interventions: Other: Follow-up of BCR TKA
- BCS TKA (Other): Patients with an afunctional or absent ACL and/or PCL will be treated with the BCS design
  Interventions: Other: Follow-up of BCS TKA
- PS TKA (Other): Patients with an afunctional or absent ACL and/or PCL will be treated with the PS design
  Interventions: Other: Follow-up of PS TKA

INTERVENTIONS:
Other: Follow-up of BCR TKA — Pre- and postoperative follow-up of patients treated with the BCR design by measuring PROMs, and clinical- and radiographic evaluation
  Other Names: Journey XR®
  Arms: BCR TKA
Other: Follow-up of BCS TKA — Pre- and postoperative follow-up of patients treated with the BCS design by measuring PROMs, and clinical- and radiographic evaluation
  Other Names: Journey BCS®
  Arms: BCS TKA
Other: Follow-up of PS TKA — Pre- and postoperative follow-up of patients treated with the PS design by measuring PROMs, and clinical- and radiographic evaluation
  Other Names: Legion PS®
  Arms: PS TKA

SUMMARY:
Today, primary total knee arthroplasty (TKA) is considered to be a safe and successful therapy for end-stage osteoarthritis of the knee. In the past decades, different total knee prostheses have been released on the market showing minor or more important differences in design features.

Smith and Nephew® (Memphis, Tennessee, USA) introduced a new posterior sacrificing (PS) design in 2005, which was called Journey BCS®, a bicruciate stabilizing design throughout knee flexion. This second generation guided motion total knee system prevents not only tibial posterior translation, but also limits tibial anterior translations by articulation between post and femoral box. As a consequence of the good results in the older population group, an increasing amount of younger and more active patients receiving TKA can be observed. In general, this age group scores remarkable lower in satisfaction. A possible explanation is the absence of anterior cruciate ligament (ACL) in these designs, which still causes abnormal kinematics. Therefore, in a further step, the research has been focusing on preserving both cruciate ligaments within the same basic design as Journey BCS®, keeping the curvature and contour of the femoral and tibial component, as well as the joint line principles. Consequently, a bi-cruciate retaining (BCR) design was developed, preserving both the ACL and posterior cruciate ligament (PCL) vessels.

BCR TKA of Smith & Nephew, called Journey XR®, has a clear potential to result in a better functional outcome while avoiding the limitations and complications of previous other designs so that previously disappointing results of the pasts are not confirmed. As a result, patients are expected to be more capable to return to an active lifestyle with normal kinematics and proprioception of the knee. New insights in biomechanics, kinetics and proprioception in native knee and TKA make higher interest in BCR TKA inevitable. Yet, there is no prospective clinical trial available that compares Journey BCS® with Journey XR® from Smith & Nephew in regard to PROMS, functional performance including gait analysis, survival and revision rates.

DETAILED DESCRIPTION:
Today, primary total knee arthroplasty (TKA) is considered to be a safe and successful therapy for end-stage osteoarthritis of the knee. In the past decades, different total knee prostheses have been released on the market showing minor or more important differences in design features. As such, knee prostheses can differ in the level of constraint they provide. More specifically, for a few decades, two main designs were available for clinical use. First, designs that only sacrifice the anterior cruciate ligament (ACL), but retain the patient's own posterior cruciate ligament (PCL), the so-called cruciate retaining (CR) design, and secondly, designs that sacrifice the patient's ACL and PCL, the so-called posterior sacrificing (PS) design. The CR design has been considered historically as the least constrained design. The containment can be adjusted by equalizing the cavity and geometry of tibial end femoral surfaces. The PS knee design, known by the cam-post mechanism, offers more constrain, but sacrifices both cruciate ligaments. In terms of complications and outcome no difference can be found between PS and CR knee designs. However, the last decade, prosthetic research focused more and more on the preservation of both PCL and ACL, in an attempt to mimic better natural kinematic behaviour of the knee and to keep the proprioceptive function of the ACL and PCL vessels.

Smith and Nephew® (Memphis, Tennessee, USA) introduced a new PS design in 2005, which was called Journey BCS®, a bicruciate stabilizing design throughout knee flexion. This second generation guided motion total knee system prevents not only tibial posterior translation, but also limits tibial anterior translations by articulation between post and femoral box. The main purpose of this type of TKA was to achieve a more normal and natural kinematic behavior with more lateral posterior roll back, while keeping the medial side stable and preserving the normal natural joint line inclination. In particular, the medial femoral condyle is more distal than lateral condyle. There is a 3° varus joint line and the convex lateral tibial surface in sagittal plane creates a slight posterior slope. More anterior translation of the femur is seen with CR design during flexion allowing possibly little more flexion in BCS design. However, although the specific design properties of this prosthesis tended to mimic the stabilizing function of the natural cruciate ligaments much better, the patient's ACL is still sacrificed and at least its proprioceptive function is still completely lost. Mid-term results of Journey II BCS® are similar compared to other knee designs. However, the younger population group seems to end up with better scores when looking at postoperative clinical and functional results. As a consequence of the good results in the older population group, an increasing amount of younger and more active patients receiving TKA can be observed. Unfortunately, a significant part of these young patients keeps complaining of residual symptoms and pain in the knee after TKA. In general, this age group scores remarkable lower in satisfaction. A possible explanation is the absence of ACL in these designs, which still causes abnormal kinematics. Furthermore, the loss of its proprioceptive function might be a factor in the mentioned feeling of imperfection. Therefore, in a further step, the research has been focusing on preserving both cruciate ligaments within the same basic design as Journey BCS®, keeping the curvature and contour of the femoral and tibial component, as well as the joint line principles. Consequently, a bi-cruciate retaining (BCR) design was developed, preserving both the ACL and PCL vessels. Patients retain better knee kinematics, stability, proprioception and consequently better functionality and satisfaction by retaining ACL in TKA. Although the design is available on the American market for about seven years, and since 2 years also on the European market, it is still not widely used, even not by surgeons who are familiar with the other designs of the same prosthetic line. One of the reasons therefore might be the published higher rates of early revisions or poly exchange of another recent design in which both cruciate ligaments are preserved, released on the market by another prosthetic company a few years earlier.

BCR TKA of Smith & Nephew, called Journey XR®, is designed to retain both cruciate ligaments. Journey XR® design has a clear potential to result in a better functional outcome while avoiding the limitations and complications of previous other designs so that previously disappointing results of the pasts are not confirmed. As a result, patients are expected to be more capable to return to an active lifestyle with normal kinematics and proprioception of the knee. Journey XR® preserves specific features of Journey BCS®, such as asymmetric femoral condyles, 3° varus joint line and low constraint concave medial and convex lateral articular surface. In order to preserve both cruciate ligaments Journey XR® design has some adjustments, which are mentioned here. Tibial base plate design with continuous keel and anterior bridge, consists of high-quality forged Ti-6Al-4V which is less stiff. These tibial component updates were implemented to reduce the risk of bone resorption from stress shielding and to double fatigue strength compared to BCR design of another company. Fixation of tibial Journey XR® baseplate, which is provided with an asymmetrical notch to accept ACL footprint, is based on four-corner peg fixation with maximal bone coverage and good results compared to known knee designs with stem fixation. Furthermore, tibial insert lock is optimized. Previous total knee designs of Smith and Nephew® already proved very limited poly wear when using highly cross-linked polyethylene (XLPE) in combination with OXINIUM, according to VERILAST® technology. Approximately 4000 Journey XR® procedures have been done globally in the last 3 years in 10 countries, among which US, Japan, South Africa and some countries in Western EU like Belgium. Currently 21% of these cases is placed using NAVIO® or Cori robot technology but this proportion is growing. Present literature is clear that retention of ACL and PCL has significant higher satisfaction compared to TKA patients, as with partial knee arthroplasty. Moreover, last update of journey XR® design of 2017 had interesting solutions for the limitations of the mentioned previous design. Problems like tibia poly wear, tibia insert lock and implant strength were common. New insights in biomechanics, kinetics and proprioception in native knee and TKA make higher interest in BCR TKA inevitable. Yet, there is no prospective clinical trial available that compares Journey BCS® with Journey XR® and the Legion PS® design from Smith & Nephew in regard to PROMS, functional performance including gait analysis, survival and revision rates.

ELIGIBILITY:
Inclusion Criteria:

* ICF obtained
* End stage bi- or tricompartmental osteoarthritis of the knee meeting the general criteria for TKA

Exclusion Criteria:

* Inflammatory arthritis (e.g. rheumatoid arthritis).
* BMI >30 due to less accurate gait analysis.
* Extension deficit of >10° and flexion deficit of <110° of the knee.
* Varus and valgus deviations >10° of the knee
* Mental retardation, a systemic disease or decline normal health causing post-operative rehabilitation cannot take place properly.
* Suggestive musculoskeletal deformity of the lower limb or vertebral column, causing postoperative rehabilitation cannot take place properly to prevent confounding. Normal joints are defined as asymptomatic joints with normal physical examination and mild to no changes on radiographs. An exception is made for primary total hip prosthesis.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-08-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Oxford Knee Score (OKS) | Within a period of 2 years
  To assess function and pain after total knee arthroplasty
EuroQol 5D-5L (EQ5D-5L) | Within a period of 2 years
  To evaluate mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
Visual Analogue Scale (VAS) | Within a period of 2 years
  To measure acute and chronic pain
Knee Range of Motion (ROM) | Within a period of 2 years
  To measure knee extension/flexion using a goniometer
Knee Society Score (KSS) | Within a period of 2 years
  To provide a simple and objective scoring system to rate the knee and patient's functional abilities before and after total knee arthroplasty.
Forgotten Joint Score (FJS) | Within a period of 2 years
  To assess how natural the prosthesis feels after total knee arthroplasty
Radiographic evaluation | Within a period of 2 years
  To perform a standard knee radiography using X-ray (face in extension, profile max flexion, axial 30° flexion) and CT-scan for measuring the knee alignment
Knee joint function during gait | Within a period of 2 years
  To assess knee joint function through instrumented motion analysis during gait
Knee joint function during motor tasks | Within a period of 2 years
  To assess knee joint function through instrumented motion analysis during motor tasks (walking up and down hill and stairs,...)
EOS full-leg radiography | Within a period of 2 years
  To perform a full-leg radiography for measuring the knee alignment

SECONDARY OUTCOMES:
Motion analysis | Within a period of 2 years
  Patients are compared to a matched control group with a healthy natural knee, available in a database.

CONTACTS AND LOCATIONS:
Overall Officials: Hilde Vandenneucker, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No